CLINICAL TRIAL: NCT00654004
Title: Fatty Acid Oxidation Disorders & Body Weight Regulation
Brief Title: Fatty Acid Oxidation Disorders & Body Weight Regulation Grant
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Oregon State University (Other)
Responsible Party: Principal Investigator, Melanie B Gillingham, Assistant Professor, Oregon Health and Science University
Other Study IDs: DK71869; K01DK071869 (NIH)
Record Dates: First submitted 2008-04-03; First posted 2008-04-07 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Trifunctional Protein Deficiency
Keywords: trifunctional; protein; deficiency; TFP; weight; regulation
MeSH Terms: conditions — Trifunctional Protein Deficiency With Myopathy And Neuropathy; Body Weight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples. Body composition and energy expenditure data. MRI/MRS images.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects: Subjects are patients with a long-chain fatty acid oxidation disorder including CPT2, VLCAD, TFP or LCHAD deficiency.
- Controls: Subjects do not have a fatty acid oxidation disorder.

SUMMARY:
Several hormones involved in body weight regulation increase the subject's ability to burn fat for energy. The purpose of this study is to investigate how burning fat for energy may affect those hormones and body weight in children. The study will also determine if eating a diet higher in protein alters the amount of fat you burn and how these hormones control body weight.

DETAILED DESCRIPTION:
A role for mitochondrial fatty acid oxidation in the peripheral signaling cascade of leptin, adiponectin and insulin has recently been proposed from animal studies but has not been investigated in humans. Children with trifunctional protein (TFP, including deficiency of long-chain hydroxyacyl-CoA dehydrogenase) and very long-chain acyl-CoA dehydrogenase (VLCAD) deficiency, inherited disorders of long-chain fatty acid ß-oxidation, lack an ability to oxidize fatty acids for energy. They have increased levels of body fat and circulating leptin and a high incidence of obesity. Current therapy for children with these disorders is based on frequent meals and consuming a low fat, very high carbohydrate diet. Despite treatment, exercise induced rhabdomyolysis is a common complication of TFP and VLCAD deficiency that frequently leads to exercise avoidance. The effects of these genetic defects on body composition and weight regulation have not been investigated. The contribution of fatty-acid oxidation during moderate intensity exercise in children has also not been reported.

Two groups of subjects were recruited: one group of subjects had a long-chain fatty acid oxidation disorder (n=13). The other group is a group of controls (n=16). We studied peripheral signals of body weight regulation, glucose tolerance, body composition, and exercise metabolism in subjects with a long-chain fatty acid oxidation disorder compared to normal controls.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of TFP, LCHAD, CPT2 or VLCAD deficiency
* at least 7 years of age
* willingness to complete overnight admission
* generally healthy

Exclusion Criteria:

* inclusion in another research project that alters macronutrient intake
* diabetes, thyroid disease or other endocrine dysfunction that alters body composition.
* pregnancy
* anemia

Ages: 7 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects were patients with a diagnosis of mitochondrial trifunctional protein, long-chain 3-hydroxyacylCoA dehydrogenase, very long-chain acylCoA dehydrogenase or carnitine palmitoyltransferase 2 deficency. They were recruited through advertisements on the FAO support website, or physician referral. Control subjects were from the greater Portland area. They were recruited via adverstisements at OHSU.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2006-04; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie B. Gillingham, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Behrend AM, Harding CO, Shoemaker JD, Matern D, Sahn DJ, Elliot DL, Gillingham MB. Substrate oxidation and cardiac performance during exercise in disorders of long chain fatty acid oxidation. Mol Genet Metab. 2012 Jan;105(1):110-5. doi: 10.1016/j.ymgme.2011.09.030. Epub 2011 Oct 1. PMID 22030098

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with a long-chain fatty acid oxidation disorder were recruited through announcements on disease specific websites, and referrals from metabolic physicians. Controls were recruited through the OHSU website and word of mouth.
Pre-assignment Details: After a subject had completed the protocol, potential control subjects were screened for age, gender and BMI that would allow for a 1 to 1 matching study design.
Period: Overall Study
Arm/Group | Subjects | Controls
Started | 14 | 12
Completed | 13 | 12
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects | Controls | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 10 | 21
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 14 (8) | 15 (7) | 14.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
  Canada | 1 | 0 | 1
  Europe | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: An Outcome of This Study is the Difference in Percent Body Fat (%BF) Between Subjects With a Long-chain Fatty Acid Oxidation Disorder and Normal Controls.
Description: Body composition by DEXA was measured in subjects with a long-chain fatty acid oxidation disorder (n=13). Twelve age, sex and BMI matched controls and 4 heterozygotes for a long-chain fatty acid oxidation disorder were recruited who also completed body composition measures. The difference in body composition between subjects and age matched controls was compared by t-test.
Time Frame: Subjects will be compared to controls at one point in time.
Population: Study design was based on 1 to 1 matching of subjects and controls. Thirteen subjects but only 12 controls completed the protocol. We report results of 12 subjects compared to 12 matched controls.
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Subjects | Controls
Number analyzed (Participants) | 12 | 12
percentage of body fat | 31.8 (6.8) | 27.2 (9.1)

2. Secondary Outcome: The Difference in Plasma Adiponectin Levels Between Subjects With a Long-chain Fatty Acid Oxidation Disorder and Matched Controls Was Compared by T-test
Description: Fasting total adiponectin levels in ug/ml were measured in both groups (subjects with a long-chain fatty acid oxidation disorder). The differences between groups were compared with a t-test
Time Frame: Fasting total adiponectin (ug/ml)
Population: Study was designed as a one to one matching design. Thirteen subjects but only 12 controls completed the protocol. We report results of 12 subjects and 12 matched controls.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Subjects | Controls
Number analyzed (Participants) | 12 | 12
ug/ml | 17.3 (7.2) | 24.4 (13.5)

3. Primary Outcome: An Outcome of This Study is the Difference in Glucose Tolerance Between Subjects With a Long-chain Fatty Acid Oxidation Disorder and Normal Controls.
Description: Glucose tolerance was estimated by the Matsuda Index using glucose and insulin values from a standard oral glucose tolerance test. The Matsuda Index is calculated by the following formula: 10,000/ sq root of (fasting glucose mg/dl X fasting insulin in units/ml) X (mean glucose (mg/dl) X mean insulin (units/ml) and correlates with insulin sensitivity measured by the gold standard method of a hyperinsulinemic euglycemic clamp. Values of 2.5 or greater are considered insulin sensitive. Values of 2.4 or less are considered insulin resistance.
  The Matsuda Index of Insulin Sensitivity was measured in subjects with a long-chain fatty acid oxidation disorder (n=12). Twelve age, sex and BMI matched controls and 4 heterozygotes for a long-chain fatty acid oxidation disorder were recruited who also completed an oral glucose tolerance test. The difference in Mastuda Index between subjects and age matched controls was compared by t-test.
Time Frame: Subjects will be compared to controls at one point in time.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects | Controls
Number analyzed (Participants) | 12 | 12
units on a scale | 2.8 (1.8) | 3.13 (1.57)

4. Secondary Outcome: The Difference in Plasma Leptin Between Subjects With a Long-chain Fatty Acid Oxidation Disorder and Matched Controls Was Compared by T-test
Description: Fasting leptin in ng/kg fat mass were measured in both groups (subjects with a long-chain fatty acid oxidation disorder; controls). The differences between groups were compared with a t-test
Time Frame: Fasting leptin levels ng per kg of fat mass
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/kg
Arm/Group | Subjects | Controls
Number analyzed (Participants) | 12 | 12
ng/kg | 0.99 (0.8) | 0.91 (0.57)

5. Secondary Outcome: The Difference in Plasma Insulin Between Subjects With a Long-chain Fatty Acid Oxidation Disorder and Matched Controls Was Compared by T-test
Description: Fasting insulin levels in uU/ml were measured in both groups. The differences between groups were compared with a t-test
Time Frame: Fasting insulin levels uUnits/ml
Population: Study was designed as a one to one matching design. Thirteen subjects but only 12 controls completed the protocol. Samples were missing on one subject so 11 subjects were compared to 11 controls.
Measure: Mean (Standard Deviation); unit: uU/ml
Arm/Group | Subjects | Controls
Number analyzed (Participants) | 11 | 11
uU/ml | 17 (8) | 13 (5)

ADVERSE EVENTS:
Description: Adverse events were assessed during the study. No serious adverse events occurred during the study.
Arm/Group | Subjects | Controls
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

LIMITATIONS AND CAVEATS:
Trial included small number of subjects with a rare disorder of long-chain fatty acid oxidation. Subjects were predominately children and adolescents. There were some technical difficulties with recruitment and collection of all the outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No